CLINICAL TRIAL: NCT00861250
Title: Assessment of Molecular Remission by ASO-RQ-PCR Technique After Induction Treatment With Bortezomib-dexamethasone (Vel/Dex) Followed by HDT With ASCT
Brief Title: Assessment of Molecular Remission by ASO-qPCR After Bortezomib-dexamethasone (Vel/Dex) Followed by ASCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Oulu University Hospital (Other); Kuopio University Hospital (Other); Helsinki University Central Hospital (Other); Kanta-Häme Central Hospital (Other Government); Seinajoki Central Hospital (Other); Jyväskylä Central Hospital (Other); Janssen-Cilag Ltd. (Industry); Päijänne Tavastia Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R08096M; 2008-003936-38 (EudraCT Number); 26866138MMY2063 (Other Grant/Funding Number: Janssen-Cilag Ltd)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2014-12

CONDITIONS: Multiple Myeloma
Keywords: Bortezomib plus dexamethasone induction therapy; Autologous stem cell transplantation; Molecular remission
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vel/Dex (Experimental)
  Interventions: Drug: bortezomib + dexamethasone

INTERVENTIONS:
Drug: bortezomib + dexamethasone — Bortezomib 1,3mg/m2 iv days 1,4,8,11, dexamethasone 40mg/day days 1-4, 9-12 in cycles 1- 2, then bortezomib 1,3mg/m2 iv days 1,4,8,11, dexamethasone 40mg/day days 1-4 in cycles 3-4, total number of cycles is 4, followed by HDT with ASCT
  Other Names: VelcadeTM

SUMMARY:
The primary objective of this study is to determine the rate of molecular remissions (MolR) assessed by ASO-RQ-PCR technique after induction treatment with bortezomib and dexamethasone (Vel/Dex) prior to high-dose therapy with melphalan and autologous stem cell transplantation (HDT-ASCT), and after HDT-ASCT in patients with multiple myeloma.

DETAILED DESCRIPTION:
HDT-ASCT is so far considered the standard of care for younger patients with multiple myeloma (MM). Current evidence indicates that quality of response is an important prognostic factor for long-term survival in MM. There are only very few data on molecular remissions (MolR) determined by the most sensitive technique, allele-specific-oligonucleotide - real-time quantitative - polymerase chain reaction (ASO-RQ-PCR) in MM, and there are no data available on molecular responses after bortezomib-based induction therapy followed by HDT-ASCT. The main aim of this study is to determine molecular response rate after ASCT following bortezomib-based induction treatment compared to a historical control group with conventional VAD induction treatment. A sensitivity of ASO-RQ-PCR technique will be compared to immunofixation and with immunophenotyping by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma
* Age 18-65 years
* Written informed consent

Exclusion Criteria:

* WHO performance status ≥ 2, unless related to MM
* Severe cardiac dysfunction
* History of hypotension
* Serious medical or psychiatric illness
* Severe hepatic dysfunction
* Severe polyneuropathy ≥ grade 2
* Active, uncontrolled infection
* Previously treated with chemotherapy or extensive radiotherapy for MM
* Known HIV positivity
* Severe renal dysfunction with need of dialyses
* History of active cancer during past 5 years, except non-melanoma skin cancer or stage 0 cervical cancer
* Female patients who are pregnant or nursing
* Male or female patients of reproductive potential who are not practising effective means of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Molecular remission after Vel/Dex induction (4 cycles) and 3-4 months after ASCT in those patients receiving CR or nCR | Before ASCT and 3-4 months after ASCT and then with 3-4 months interval

CONTACTS AND LOCATIONS:
Overall Officials: Raija H Silvennoinen, MD, Principal Investigator — Tampere University Hospital, Kuopio University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

REFERENCES:
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/25303369 — First study article: http://www.ncbi.nlm.nih.gov/pubmed/23206270